CLINICAL TRIAL: NCT03723993
Title: Effect of Remote Ischemic Preconditioning on Serum Lactate Levels As Well As Cardiac and Renal Functions During and After Open Heart Surgeries
Brief Title: Remote Ischemic Preconditioning During Cardiopulmonary Bypass
Acronym: RIPC
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Finished
Sponsor: Fayoum University (Other)
Responsible Party: Principal Investigator, Mohamed Ahmed Hamed, Lecturer of anesthesia, Fayoum University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: R123
Record Dates: First submitted 2018-10-26; First posted 2018-10-30 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-02

CONDITIONS: Lactic Acidosis
Keywords: Ischemic preconditioning; Lactate level; Cardiopulmonary bypass
MeSH Terms: conditions — Acidosis, Lactic

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Placebo Comparator): control group will have non inflated cuff around the arm.
  Interventions: Device: Non inflated cuff
- RIPC group (Active Comparator): Inflated cuff will be done systematically and regularly
  Interventions: Device: Inflated cuff

INTERVENTIONS:
Device: Inflated cuff — After patient being draped, applying cuff inflation will be done to the upper arm not having the arterial line inserted of about 200 mmHg or 15 mmHg above patient's systolic pressure 3 cycles 5 minutes each followed by 5 minutes of pressure relieve
  Arms: RIPC group
Device: Non inflated cuff — non inflated cuff around the arm for the control group
  Arms: Control group

SUMMARY:
The objective of study is to detect effect of remote ischemic preconditioning on serum lactate levels during and after cardiac surgery with cardiopulmonary bypass in addition to its effect on cardiac and renal clinical outcomes.

DETAILED DESCRIPTION:
Remote ischemic preconditioning (RIPC) is a phenomenon where transient non-injurious ischemia/ reperfusion episodes applied to an organ away from the heart can protect the myocardium from ischemia/reperfusion injury. RIPC has been found to be an attractive strategy to reduce myocardial injury and improve outcome in patients undergoing cardiac surgery. The exact mechanisms of this protection are not yet known, although stimulation of prosurvival intracellular kinase responses and inhibition of inflammatory pathways each play a role.

RIPC can be performed by noninvasive inflation and deflation of a standard blood pressure cuff or pneumatic tourniquet on the upper or lower limbs to induce brief ischemia and reperfusion, which is the mechanism by which injury in patients undergoing open cardiac surgery occurs.

ANESTHETIC TECHNIQUE All patients will be preoperatively examined and investigated by complete blood count, coagulation profile, renal and kidney functions and electrolytes. Electrocardiography, chest x ray and echocardiography will be routinely done. Coronary angiography and carotid arterial duplex will be requested in patients prepared for coronary artery bypass graft (CABG).

Patient will be premedicated by intramuscular injection of 10mg morphine in the morning of the operation. Before induction of anesthesia, a five-lead electrocardiography system will be applied to monitor heart rate, rhythm, and ST segments (leads II and V5). A pulse oximeter probe will be attached, and a peripheral venous cannula will be placed. For measurement of arterial pressure and blood sampling, a 20 G cannula will be inserted into either right or left radial artery under local anesthesia. General anesthesia will be induced by fentanyl (3-5 μg/kg), propofol titrated according to response, followed by atracurium (0.5 mg/kg).

Trachea will be intubated, patients will be mechanically ventilated with oxygen in air so as to achieve normocarbia. This will be confirmed by radial arterial blood gas analysis. An esophageal temperature probe and a Foley catheter will also be placed.

For drug infusion, a triple-lumen central venous catheter will be inserted via the right internal jugular vein.

Anesthesia will be maintained by inhaled isoflurane, with additional fentanyl injected prior to skin incision as well as sternotomy and atracurium infusion for continued muscle relaxation.

During extracorporeal circulation, patients will receive propofol infusion in addition to atracurium infusion.

Before initiation of cardiopulmonary bypass (CPB), the patients will receive intravenously tranexamic acid (2 g) and heparin (300-500 units/kg body weight) to achieve an activated clotting time > 400 s. CPB was instituted via an ascending aortic cannula and a two-stage right atrial cannula. Before, during, and after CPB (pump blood flow: 2.4 l/min/m2), mean arterial pressure was adjusted to exceed 60 mmHg. Cardiac arrest will be induced with cold antegrade crystalloid cardioplegia (St Thomas solution) or warm intermittent antegrade blood cardioplegia. Lactate-enriched Ringer's solution will be added to the CPB circuit to maintain reservoir volume when needed, and packed red blood cells will be added when hemoglobin concentration decrease to less than 7 g/dl.

After rewarming the patient to 37°C and separation from CPB, reversal of heparin by protamine sulfate, and sternal closure, the patients will be transferred to the intensive care unit.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age or older
* Elective cardiovascular surgery requiring cardiopulmonary bypass either for CABG or valve replacement.

Exclusion Criteria:

* Patients with emergency surgeries.
* Off pump heart surgery.
* Hepatic affection (INR>2).
* Renal affection (creatinine >1.6 mg/dl for men and >1.4 mg/dl for women).
* Peripheral vascular disease affecting upper limbs.
* Patients taking the antidiabetic sulphonylurea glyburide ( glibenclamide) or receiving nicorandil drug therapy will be excluded because these agents have been shown to abolish preconditioning.
* Patients being considered for radial artery conduit harvesting.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2018-11-15 (Estimated); Study Completion 2018-12-15 (Estimated)

PRIMARY OUTCOMES:
Serum lactate level | 1 minute at the end of operation
  mmol/l from arterial blood gas sample

SECONDARY OUTCOMES:
Serum lactate level | 3 minutes after induction of anesthesia
  mmol/l from arterial blood gas sample
Serum lactate level | 30 minutes, after cardiopulmonary bypass
  mmol/l from arterial blood gas sample
Serum lactate level | 1 minute before cardiopulmonary bypass
  mmol/l from arterial blood gas sample
Serum lactate level | 24 hours postoperatively.
  mmol/l from arterial blood gas sample
Serum lactate level | 48 hours postoperatively.
  mmol/l from arterial blood gas sample
Serum lactate level | 72 hours postoperatively.
  mmol/l from arterial blood gas sample
Heart rate | 2 minutes before induction of general anesthesia
  beat per minute from electrocardiogram
Heart rate | 3 minutes after induction of general anesthesia
  beat per minute from electrocardiogram
Heart rate | Every 30 minutes for 6 hours during surgery except at cardiopulmonary bypass as there is cardioplegia
  beat per minute from electrocardiogram
Systolic blood pressure | 2 minutes before induction of general anesthesia
  Measured by mmHg from invasive arterial blood pressure
Systolic blood pressure | 3 minutes after induction
  Measured by mmHg from invasive arterial blood pressure
Systolic blood pressure | Every 30 minutes for 6 hours during surgery except at cardiopulmonary bypass as there is cardioplegia and no pulsatile blood pressure
  Measured by mmHg from invasive arterial blood pressure
Diastolic blood pressure | 2 minutes before induction of general anesthesia
  Measured by mmHg from invasive arterial blood pressure
Diastolic blood pressure | 3 minutes after induction
  Measured by mmHg from invasive arterial blood pressure
Diastolic blood pressure | Every 30 minutes for 6 hours during surgery except at cardiopulmonary bypass as there is cardioplegia and no pulsatile blood pressure
  Measured by mmHg from invasive arterial blood pressure
Left ventricular fractional shortening (LVFS) | 12 hours before the operation
  measured in percentage derived from echocardiography
Left ventricular fractional shortening (LVFS) | 2 hours after the operation
  measured in percentage derived from echocardiography
Left ventricular fractional shortening (LVFS) | 4 hours after the operation
  measured in percentage derived from echocardiography
Left ventricular fractional shortening (LVFS) | 12 hours after the operation
  measured in percentage derived from echocardiography
Left ventricular fractional shortening (LVFS) | 24 hours after the operation
  measured in percentage derived from echocardiography
Left ventricular fractional shortening (LVFS) | 48 hours after the operation
  measured in percentage derived from echocardiography
Left ventricular fractional shortening (LVFS) | 72 hours after the operation
  measured in percentage derived from echocardiography
Left ventricular ejection fraction (LVEF) | 12 hours before the operation
  measured in percentage derived from echocardiography
Left ventricular ejection fraction (LVEF) | 2 hours after the operation
  measured in percentage derived from echocardiography
Left ventricular ejection fraction (LVEF) | 4 hours after the operation
  measured in percentage derived from echocardiography
Left ventricular ejection fraction (LVEF) | 12 hours after the operation
  measured in percentage derived from echocardiography
Left ventricular ejection fraction (LVEF) | 24 hours after the operation
  measured in percentage derived from echocardiography
Left ventricular ejection fraction (LVEF) | 48 hours after the operation
  measured in percentage derived from echocardiography
Central venous pressure | Baseline 2 minutes after insertion of central venous catheter
  from central venous catheter measured in cm H2O
Central venous pressure | 2 minutes before cardiopulmonary bypass
  from central venous catheter measured in cm H2O
Central venous pressure | 2 minutes after cardiopulmonary bypass
  from central venous catheter measured in cm H2O
Central venous pressure | 1 minute after the end of operation
  from central venous catheter measured in cm H2O
Serum urea level | 5 minutes before beginning of operation
  mmol/L
Serum urea level | 5 minutes after ICU admission
  mmol/L
Serum creatinine level | 5 minutes before beginning of operation
  mmol/L
Serum creatinine level | 24 hours postoperatively
  mmol/L
Serum creatinine level | 48 hours postoperatively
  mmol/L
Serum creatinine level | 72 hours postoperatively
  mmol/L
Acute kidney injury (AKI) score | 24 hours postoperatively
  Grade 1: serum creatinine rise of 150%-200% of baseline and/or urine output <0.5 mL/kg/h for >6 contiguous hours.
  Grade 2: serum creatinine rise of 200%-300% of baseline and/or urine output <0.5 mL/kg/h for >12 contiguous hours.
  Grade 3: serum creatinine rise of >300% of baseline and/or urine output <0.3 mL/kg/h for >24 h or anuria for 12 h.
Acute kidney injury (AKI) score | 48 hours postoperatively
  Grade 1: serum creatinine rise of 150%-200% of baseline and/or urine output <0.5 mL/kg/h for >6 contiguous hours.
  Grade 2: serum creatinine rise of 200%-300% of baseline and/or urine output <0.5 mL/kg/h for >12 contiguous hours.
  Grade 3: serum creatinine rise of >300% of baseline and/or urine output <0.3 mL/kg/h for >24 h or anuria for 12 h.
Acute kidney injury (AKI) score | 72 hours postoperatively
  Grade 1: serum creatinine rise of 150%-200% of baseline and/or urine output <0.5 mL/kg/h for >6 contiguous hours.
  Grade 2: serum creatinine rise of 200%-300% of baseline and/or urine output <0.5 mL/kg/h for >12 contiguous hours.
  Grade 3: serum creatinine rise of >300% of baseline and/or urine output <0.3 mL/kg/h for >24 h or anuria for 12 h.
Serum sodium level | 5 minutes after ICU admission.
  milliequivalent/L
Serum sodium level | 5 minutes before beginning of operation
  milliequivalent/L
Serum potassium level | 5 minutes before beginning of operation
  milliequivalent/L
Serum potassium level | 5 minutes after ICU admission
  milliequivalent/L
Arterial oxygen pressure | 5 minutes before operation
  From arterial blood gas sampling
Arterial oxygen pressure | 2 minutes before cardiopulmonary bypass
  From arterial blood gas sampling
Arterial oxygen pressure | 2 minutes after cardiopulmonary bypass
  From arterial blood gas sampling
Arterial oxygen pressure | 1 minute after end of operation
  From arterial blood gas sampling
Arterial oxygen pressure | Every 6 hours for 24 hours in the ICU
  From arterial blood gas sampling
Arterial carbon dioxide pressure | 5 minutes before operation
  From arterial blood gas sampling
Arterial carbon dioxide pressure | 2 minutes before cardiopulmonary bypass
  From arterial blood gas sampling
Arterial carbon dioxide pressure | 2 minutes after cardiopulmonary bypass
  From arterial blood gas sampling
Arterial carbon dioxide pressure | 1 minute after end of operation
  From arterial blood gas sampling
Arterial carbon dioxide pressure | Every 6 hours for 24 hours in the ICU
  From arterial blood gas sampling
Power of hydrogen (pH) | 5 minutes before operation
  From arterial blood gas sampling
Power of hydrogen (pH) | 2 minutes before cardiopulmonary bypass
  From arterial blood gas sampling
Power of hydrogen (pH) | 2 minutes after cardiopulmonary bypass
  From arterial blood gas sampling
Power of hydrogen (pH) | 1 minute after end of operation
  From arterial blood gas sampling
Power of hydrogen (pH) | Every 6 hours for 24 hours in the ICU
  From arterial blood gas sampling
Standard bicarbonate level | 5 minutes before operation
  From arterial blood gas sampling
Standard bicarbonate level | 2 minutes before cardiopulmonary bypass
  From arterial blood gas sampling
Standard bicarbonate level | 2 minutes after cardiopulmonary bypass
  From arterial blood gas sampling
Standard bicarbonate level | 1 minute after end of operation
  From arterial blood gas sampling
Standard bicarbonate level | Every 6 hours for 24 hours in the ICU
  From arterial blood gas sampling

OTHER OUTCOMES:
Age | 1 hour before operation once the patient is recruited
  in years

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed A Hamed, MD, Principal Investigator — Faculty of medicine, Fayoum University
Locations (1):
- Mohamed Hamed, Al Fayyum, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Saxena P, Newman MA, Shehatha JS, Redington AN, Konstantinov IE. Remote ischemic conditioning: evolution of the concept, mechanisms, and clinical application. J Card Surg. 2010 Jan-Feb;25(1):127-34. doi: 10.1111/j.1540-8191.2009.00820.x. Epub 2009 Jun 22. PMID 19549044
- [Background] Heusch G. Cardioprotection: chances and challenges of its translation to the clinic. Lancet. 2013 Jan 12;381(9861):166-75. doi: 10.1016/S0140-6736(12)60916-7. Epub 2012 Oct 22. PMID 23095318
- [Background] Thielmann M, Kottenberg E, Kleinbongard P, Wendt D, Gedik N, Pasa S, Price V, Tsagakis K, Neuhauser M, Peters J, Jakob H, Heusch G. Cardioprotective and prognostic effects of remote ischaemic preconditioning in patients undergoing coronary artery bypass surgery: a single-centre randomised, double-blind, controlled trial. Lancet. 2013 Aug 17;382(9892):597-604. doi: 10.1016/S0140-6736(13)61450-6. PMID 23953384
- [Background] Badreldin AM, Doerr F, Elsobky S, Brehm BR, Abul-dahab M, Lehmann T, Bayer O, Wahlers T, Hekmat K. Mortality prediction after cardiac surgery: blood lactate is indispensible. Thorac Cardiovasc Surg. 2013 Dec;61(8):708-17. doi: 10.1055/s-0032-1324796. Epub 2013 Mar 11. PMID 24338631